CLINICAL TRIAL: NCT02049359
Title: Use of a Short Messaging Service for Optimizing Hemoglobin A1C Management in Low-Income Diabetic Patients (SAMI TRIAL)
Brief Title: Short Messaging Service for Optimizing Hemoglobin A1C Management in Low-Income Diabetics
Acronym: SAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell University, Incorporated (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Care as usual; no bidirectional texting
- Texting (Experimental): Bidirectional texting weekly for 12 weeks
  Interventions: Other: Texting

INTERVENTIONS:
Other: Texting — Bidirectional texting once weekly for 12 weeks
  Arms: Texting

SUMMARY:
The purpose of this study is to determine the impact of two-way short message service (SMS) on glycemic control in low-income, poorly-controlled adult diabetic patients.

DETAILED DESCRIPTION:
This multi-center, unblinded, prospective randomized controlled trial will enroll adult diabetic patients of the Wilson Community Health Center, Harvest Family Health Center, and Freedom Hill Community Health Center living below 200% of 2013 poverty level with a serum hemoglobin A1C >9% and who currently own a mobile device with text messaging capacity. After written informed consent has been obtained, subjects will be randomized to intervention or control group (1:1), stratified based on insulin initiation within 1 week of study inclusion. Participants randomized to the intervention group will be further divided into subgroups as "insulin user" or "non-insulin user" and both will receive SMS messages every 7 days. The content of the message consist of medication reminders, reporting of blood glucose results, insulin technique assessment (if applicable), or d) medication adherence assessment. Participants will be asked to respond with a simple text within 7 days. The intervention group will receive the standard medical appointment reminder via telephone one to two business days prior to the appointment at the Health Center PLUS a unidirectional text message two business days prior to scheduled health center appointments. Control group participants will receive the standard medical appointment reminder via telephone one to two business days prior to the appointment at the health center. All participants in the study (control and intervention) will undergo venipuncture at 3 months (+/-) 2 weeks for the determination of hemoglobin A1C. Demographic information, and frequency of hemoglobin A1C concentrations in the past 6 months will be assessed at baseline. Each week for 12 weeks, the number of texts sent per week and by type, percent of respondents weekly by text or by phone, content of participant responses, number of patients unable to be reached via text, total investigator time spent per week, and time spent per contact will be recorded. At the three month visit, the hemoglobin A1C concentration, blood transfusions since study initiation, and medication changes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* New or existing patient of Carolina Family Health Centers Inc. (Wilson Community Health Center, Harvest Family Health Center, Freedom Hill Community Health Center)
* Diagnosis of diabetes
* Single serum hemoglobin A1C equal to or greater than 9% within 2 weeks of study enrollment
* Below 200% of 2013 poverty level
* Currently own a mobile device with text messaging capacity and anticipated service for duration of 12 week study period

Exclusion Criteria:

* Anemia diagnosed within past 3 months
* Blood transfusion within the past 3 months
* unable to read English at the fifth grade level

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Smith, PharmD, Principal Investigator — Campbell University/Wilson Community Health Center; Richard Drew, PharmD, Study Director — Campbell University/Duke University
Locations (3):
- United States (3):
  - Harvest Family Health Center, Elm City, North Carolina
  - Freedom Hill Community Health Center, Tarboro, North Carolina
  - Wilson Community Health Center, Wilson, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Texting
Started | 95 | 75
Completed | 69 | 56
Not Completed | 26 | 19
Not completed — Lost to Follow-up | 26 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Texting | Total
Number analyzed (Participants) | 69 | 56 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 51 | 116
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.7) | 52.5 (10.3) | 51.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 32 | 73
  Male | 28 | 24 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 50 | 42 | 92
  Caucasian | 15 | 10 | 25
  Hispanic | 2 | 1 | 3
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 56 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline A1C
Description: Change in A1C from baseline
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of A1C decrease
Arm/Group | Control Group | Texting
Number analyzed (Participants) | 69 | 56
percentage of A1C decrease | 1.1 [0.6 to 1.6] | 1.4 [0.9 to 1.8]

2. Secondary Outcome: Change in A1C Based on Age, Gender, Race, Type and Duration of Diabetes
Description: Change in A1C from baseline based on age, gender, race, type and duration of diabetes
Time Frame: 12 weeks
Population: Change in A1C percentage from baseline by demographic characteristics
Measure: Mean (95% Confidence Interval); unit: percentage of A1C decrease
Arm/Group | Control Group | Texting
Number analyzed (Participants) | 69 | 56
percentage of A1C decrease
  Age 18-35: number analyzed (Participants) | 7 | 5
  Age 18-35 | 2.1 [0.3 to 4.0] | 1.9 [0.5 to 2.0]
  36-55 years: number analyzed (Participants) | 32 | 29
  36-55 years | 1.2 [0.5 to 1.8] | 1.4 [0.8 to 2.1]
  56-65 years: number analyzed (Participants) | 26 | 17
  56-65 years | 0.5 [0.2 to 1.2] | 1.5 [0.5 to 2.6]
  >65 years: number analyzed (Participants) | 4 | 5
  >65 years | 0.8 [0.33 to 1.9] | 1.2 [0.2 to 2.2]
  African American: number analyzed (Participants) | 50 | 42
  African American | 1.2 [0.5 to 1.7] | 1.3 [0.7 to 1.8]
  Caucasian: number analyzed (Participants) | 15 | 10
  Caucasian | 1.0 [0.2 to 1.7] | 1.4 [0.8 to 2.0]
  Hispanic: number analyzed (Participants) | 2 | 1
  Hispanic | 2.0 [NA to NA] — Sample inadequate to describe 95% confidence intervals | 0.9 [NA to NA] — Sample inadequate to describe 95% confidence intervals
  Other: number analyzed (Participants) | 2 | 3
  Other | 1.0 [NA to NA] — Sample inadequate to describe 95% confidence intervals | 3.0 [NA to NA] — Sample inadequate to describe 95% confidence intervals
  Female: number analyzed (Participants) | 41 | 32
  Female | 0.9 [0.3 to 1.4] | 1.3 [0.8 to 1.7]
  Male: number analyzed (Participants) | 28 | 24
  Male | 1.4 [0.6 to 2.4] | 1.5 [0.7 to 2.4]

ADVERSE EVENTS:
Arm/Group | Control Group | Texting
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/75
Other Adverse Events (participants affected / at risk) | 0/95 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes